CLINICAL TRIAL: NCT01578031
Title: Responses to CPAP Treatment in Obese and Lean Sleep Apnea Patients
Brief Title: The Effects of Treating Obese and Lean Patients With Sleep Apnea
Acronym: PISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIH P02 HL094307-01
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Sleep Apnea; Obesity
Keywords: Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Obese Patients with Obstructive Sleep Apnea (Active Comparator): Obese adults between the 40 and 65 years of age with a new diagnosis of OSA as evidenced by an apnea/hypopnea index ≥ 15, ≤ 75 episodes per hour, who are naïve to CPAP use will be started on CPAP treatment.
  Interventions: Device: Positive Airway Pressure During Sleep (ResMed S9 Elite)
- Non-obese Patients with Obstructive Sleep Apnea (Active Comparator): Non-obese adults between the 40 and 65 years of age with a new diagnosis of OSA as evidenced by an apnea/hypopnea index ≥ 15, ≤ 75 episodes per hour, who are naïve to CPAP use will be started on CPAP treatment.
  Interventions: Device: Positive Airway Pressure During Sleep (ResMed S9 Elite)
- Obese subjects without OSA (Other): Control.
  Interventions: Other: Usual Care
- Non-obese subjects without OSA (Other): Control.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Positive Airway Pressure During Sleep (ResMed S9 Elite) — Positive airway pressure during sleep (ResMed S9 Elite).
  Arms: Non-obese Patients with Obstructive Sleep Apnea; Obese Patients with Obstructive Sleep Apnea
Other: Usual Care — Usual care.
  Arms: Non-obese subjects without OSA; Obese subjects without OSA

SUMMARY:
The investigators' overall goal is to compare the effect of CPAP treatment on intermediate cardiovascular risk measures in obese versus lean patients with obstructive sleep apnea (OSA). The overall hypothesis is that, adjusting for OSA severity and obtaining normative data from non-OSA subjects with comparable amounts of visceral adiposity, the two OSA groups will have comparable improvements in daytime sleepiness, but that the cardiovascular and metabolic improvements following CPAP therapy will be decreased in OSA patients with increased visceral adipose tissue. The investigators anticipate that, although there will be a greater absolute change in markers of sympathetic activity, inflammation and oxidative stress in obese compared to lean OSA patients following CPAP treatment, the levels will still be abnormally high in the obese patients resulting in the decreased improvements in insulin resistance, arterial blood pressure, and vascular health in obese versus lean OSA patients.

DETAILED DESCRIPTION:
Obesity and obstructive sleep apnea (OSA) are independent risk factors for insulin resistance, systemic hypertension and cardiovascular disease. Both obesity and OSA are associated with increased sympathetic activity, inflammatory activity, and oxidative stress, the presumed mediators of their shared clinical consequences. Due to the conflicting results of previous intervention studies treating OSA patients with CPAP, the investigators still do not know if treatment of obese OSA patients has a substantial benefit on these risk factors. In Aim 1, to determine the effects of obesity on the response to CPAP treatment in OSA patients, the investigators will compare responses in daytime sleepiness, insulin resistance, and arterial blood pressure following CPAP treatment in obese and lean OSA patients, stratified by the amount of abdominal visceral adipose tissue, a fat depot associated with increased sympathetic activity, inflammation, and oxidative stress, and a more powerful predictor than BMI of adverse cardiovascular and metabolic outcomes. Aim 2 will determine the effect of CPAP treatment in these two patients groups on sympathetic activity, and inflammatory and oxidative stress biomarkers. The overall hypothesis is that, adjusting for OSA severity and obtaining normative data from non-OSA subjects with comparable amounts of visceral adiposity (Aim 3), the two OSA groups will have comparable improvements in daytime sleepiness, but that the cardiovascular and metabolic improvements following CPAP therapy will be decreased in OSA patients with increased visceral adipose tissue. The investigators anticipate that, although there will be a greater absolute change in markers of sympathetic activity, inflammation and oxidative stress in obese compared to lean OSA patients following CPAP treatment, the levels will still be abnormally high in the obese patients resulting in the decreased improvements in insulin resistance, arterial blood pressure, and vascular health in obese versus lean OSA patients. Relevance: Obese patients are at increased risk of developing sleep apnea. Both obesity and sleep apnea are felt to increase the risk of diabetes, hypertension, and cardiovascular disease. The proposed research will begin to determine if treating obese patients with sleep apnea helps to reduce these risks. If the beneficial effects of CPAP treatment are reduced in obese compared to lean patients with sleep apnea, then treatment of sleep apnea in obese patients needs to be combined with effective management of their obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 years; Will only recruit post-menopausal women not on hormone replacement therapy to avoid the potential confounding effects of female hormones on OSA prevalence and severity, fat distribution as well as the end-points (50-60)
* Lean subjects need to have a waist circumference score <= 107 cm in men and <= 96 cm in women.
* Obese subjects need to have a waist circumference score > 107 cm in men and > 96 cm in women
* For OSA volunteers, 15 ≤ AHI ≤ 75 (see Preliminary Results for justification of upper limit) on full-night in-laboratory polysomnogram within the last 6 months.
* Stable medical history and no change in medications, including anti-hypertensive and lipid-lowering medications, in the previous 2 months
* No regular daytime use (> 3 times/week) of sedative or hypnotic medications in the last 2 months
* Arm circumference ≤ 50 cm (manufacturer limit for performing ambulatory BP recording)

Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Not satisfied with reimbursement
* Time constraints
* No telephone access or inability to return for follow up testing.
* BMI > 40 kg/m2.
* Diagnosis of another sleep disorder in addition to OSA based on PSG (e.g., periodic limb movement disorder [≥ 15 limb movements/hour of sleep with arousal], central sleep apnea [≥ 50% of apneas on diagnostic PSG are central apneas], insomnia, restless legs syndrome obesity hypoventilation syndrome, or narcolepsy).
* Previous treatment with positive airway pressure, home oxygen therapy, tracheotomy, uvulopalatopharyngoplasty, or other surgery for OSA
* Requiring oxygen or bi-level positive airway pressure for treatment of OSA.
* A clinically unstable medical condition as defined by a new diagnosis or change in medical management in the previous 2 months (e.g., myocardial infarction, congestive heart failure, Cheyne-Stokes breathing, unstable angina, thyroid disease, depression or psychosis, ventricular arrhythmias, cirrhosis, surgery, or recently diagnosed cancer)
* Positive urine toxicology screen
* Rotating Night shift workers in situations or occupations where they regularly experience jet lag, or have irregular work schedules by history over the last 6 months.
* Routine consumption of more than 2 alcoholic beverages per day as determined by the CAGE questionnaire (63-65).
* Unable to perform tests due to inability to communicate verbally, inability to write and read in English; less than a 5th grade reading level; visual, hearing or cognitive impairment (e.g. previous head injury); or upper extremity motor deficit (e.g., previous stroke that prevents patient from using CPAP treatment).
* Current illicit drug use
* Excessive caffeine use (More than 10 caffeinated beverages per day)
* Recent or recurring history of recreational drug use leading to tolerance or dependance.
* Subjects with known moderate to severe renal disease will not undergo the enhanced or dynamic portion of the study.
* Women with a positive pregnancy test will be excluded from the study.
* Subjects who are found to have mild sleep apnea will be ineligible to participate further in the study and will paid up until that time.
* Active infection, malignancy or chronic inflammatory disorders such as autoimmune diseases since these conditions can alter inflammatory biomarker levels.
* No metal parts in the body as participants would not be allowed to enter the magnet during their MRI

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kuna, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Imayama I, Gupta A, Yen PS, Chen YF, Keenan B, Townsend RR, Chirinos JA, Weaver FM, Carley DW, Kuna ST, Prasad B. Socioeconomic status impacts blood pressure response to positive airway pressure treatment. J Clin Sleep Med. 2022 May 1;18(5):1287-1295. doi: 10.5664/jcsm.9844. PMID 34931603
- [Derived] Xu L, Keenan BT, Maislin D, Gislason T, Benediktsdottir B, Gudmundsdottir S, Gardarsdottir M, Staley B, Pack FM, Guo X, Feng Y, Chahwala J, Manaktala P, Hussein A, Reddy-Koppula M, Hashmath Z, Lee J, Townsend RR, Schwab RJ, Pack AI, Kuna ST, Chirinos JA. Effect of Obstructive Sleep Apnea and Positive Airway Pressure Therapy on Cardiac Remodeling as Assessed by Cardiac Biomarker and Magnetic Resonance Imaging in Nonobese and Obese Adults. Hypertension. 2021 Mar 3;77(3):980-992. doi: 10.1161/HYPERTENSIONAHA.120.15882. Epub 2021 Jan 19. PMID 33461313
- [Derived] Feng Y, Maislin D, Keenan BT, Gislason T, Arnardottir ES, Benediktsdottir B, Chirinos JA, Townsend RR, Staley B, Pack FM, Sifferman A, Pack AI, Kuna ST. Physical Activity Following Positive Airway Pressure Treatment in Adults With and Without Obesity and With Moderate-Severe Obstructive Sleep Apnea. J Clin Sleep Med. 2018 Oct 15;14(10):1705-1715. doi: 10.5664/jcsm.7378. PMID 30353806

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants enrolled is the number of participants who agreed to participate in the study following completion of the informed consent process. The number of participants Started is the number of participants who were assigned to each Arm/Group.
Period: Overall Study
Arm/Group | Obese Patients With Obstructive Sleep Apnea | Non-obese Patients With Obstructive Sleep Apnea | Obese Subjects Without OSA | Non-obese Subjects Without OSA
Started | 129 | 69 | 12 | 30
Completed | 67 (Follow-up obtained only in subjects with average PAP use at least 4 hr/day) | 35 (Follow-up obtained only in subjects with average PAP use at least 4 hr/day) | 12 (Only baseline data collected) | 30 (Only baseline data collected)
Not Completed | 62 | 34 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Patients With Obstructive Sleep Apnea | Non-obese Patients With Obstructive Sleep Apnea | Obese Subjects Without OSA | Non-obese Subjects Without OSA | Total
Number analyzed (Participants) | 129 | 69 | 12 | 30 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 129 | 69 | 12 | 30 | 240
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (7.1) | 52.7 (6.5) | 54.3 (7.8) | 51.8 (5.8) | 53.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 2 | 6 | 41
  Male | 106 | 59 | 10 | 24 | 199
Region of Enrollment [Number; unit: participants]
  United States | 71 | 27 | 3 | 15 | 116
  Iceland | 58 | 42 | 9 | 15 | 124

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Arterial Blood Pressure
Description: Change in mean 24-hour ambulatory blood pressure from baseline following 4-months of PAP treatment
Time Frame: 4 months
Population: These numbers reflect the overall number of participants who completed 4 months of CPAP treatment (i.e., the completer's analysis) and have complete data for this outcome.
Measure: Mean (Inter-Quartile Range); unit: mm Hg
Arm/Group | Obese Patients With Obstructive Sleep Apnea | Non-obese Patients With Obstructive Sleep Apnea
Number analyzed (Participants) | 88 | 46
mm Hg | -4.21 [-7.12 to -1.29] | -0.95 [-4.02 to 2.12]

2. Secondary Outcome: Change From Baseline in Psychomotor Vigilance Task
Description: Change from Baseline in Psychomotor Vigilance Task as measured by number of lapses during 10-minute Reaction time test.
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lapses
Arm/Group | Obese Patients With Obstructive Sleep Apnea | Non-obese Patients With Obstructive Sleep Apnea
Number analyzed (Participants) | 92 | 50
lapses | -0.27174 (2.19) | -0.7778 (2.47)

3. Secondary Outcome: Change From Baseline in Sympathetic Nervous System Activity
Description: Change from Baseline in Sympathetic Nervous System Activity as measured by 24-hour urine collection for norepinephrine levels.
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/24 hours
Arm/Group | Obese Patients With Obstructive Sleep Apnea | Non-obese Patients With Obstructive Sleep Apnea
Number analyzed (Participants) | 104 | 55
mcg/24 hours | -5.9011 (9.4996) | -3.0649 (11.987)

4. Secondary Outcome: Change From Baseline in Circulating Inflammatory Biomarker
Description: Change from Baseline in Circulating Inflammatory Biomarker: IL-6.
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Obese Patients With Obstructive Sleep Apnea | Non-obese Patients With Obstructive Sleep Apnea
Number analyzed (Participants) | 106 | 54
pg/mL | 0.153 (1.82) | -0.0211 (1.7)

5. Secondary Outcome: Change From Baseline in Oxidative Stress
Description: Overnight urinary excretion of 8-isoprostane.
Time Frame: 4 months
Population: Data were not collected.
Arm/Group | Obese Patients With Obstructive Sleep Apnea | Non-obese Patients With Obstructive Sleep Apnea
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment until completion of tests and procedures
Groups:
- Obese Patients Without Sleep Apnea: Control Obese adults between the 40 and 65 years of age without OSA as evidenced by an apnea/hypopnea index < 15
- Non-obese Patients Without Sleep Apnea: Control Non-obese adults between the 40 and 65 years of age without OSA as evidenced by an apnea/hypopnea index < 15
Arm/Group | Obese Patients With Obstructive Sleep Apnea | Non-obese Patients With Obstructive Sleep Apnea | Obese Patients Without Sleep Apnea | Non-obese Patients Without Sleep Apnea
All-Cause Mortality (participants affected / at risk) | 1/129 | 0/69 | 0/12 | 0/30
Serious Adverse Events (participants affected / at risk) | 5/129 | 4/69 | 0/12 | 0/30
Other Adverse Events (participants affected / at risk) | 32/129 | 7/69 | 3/12 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obese Patients With Obstructive Sleep Apnea (N=129) | Non-obese Patients With Obstructive Sleep Apnea (N=69) | Obese Patients Without Sleep Apnea (N=12) | Non-obese Patients Without Sleep Apnea (N=30)
Hospitalization (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hospitalization (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hospitalizaiton (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obese Patients With Obstructive Sleep Apnea (N=129) | Non-obese Patients With Obstructive Sleep Apnea (N=69) | Obese Patients Without Sleep Apnea (N=12) | Non-obese Patients Without Sleep Apnea (N=30)
High blood pressure (Cardiac disorders) | 11 (11) | 7 (7) | 3 (3) | 0 (0)
Claustrophobia during MRI (Psychiatric disorders) | 10 (10) | 0 (0) | 1 (1) | 0 (0)
Abnormal finding on MiniScid (Psychiatric disorders) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Abnormal MRI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal spirometry (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No